CLINICAL TRIAL: NCT00575185
Title: Randomized, Placebo-Controlled, Double-Blind Study to Assess Clinical and Antiviral Activity of Valomaciclovir (EPB 348) in Infectious Mononucleosis Due to Primary Epstein-Barr Virus Infection (Mono 6)
Brief Title: Activity of Valomaciclovir in Infectious Mononucleosis Due to Primary Epstein-Barr Virus Infection
Acronym: Mono6
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Epiphany Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0709M16341
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Infectious Mononucleosis
Keywords: Mono; Mononucleosis; Epstein-Barr virus
MeSH Terms: conditions — Infectious Mononucleosis; Epstein-Barr Virus Infections | interventions — valomaciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valomaciclovir (Active Comparator): Valomaciclovir 2 grams orally twice daily for 21 days
  Interventions: Drug: Valomaciclovir
- placebo (Placebo Comparator): placebo 2 tablets twice daily for 21 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Valomaciclovir — 4 grams orally of valomaciclovir (2 grams BID) for 21 days.
  Arms: Valomaciclovir
Drug: placebo — Placebo tablets orally twice daily for 21 days.
  Arms: placebo

SUMMARY:
This will be a randomized, placebo-controlled, double-blind single-center proof of concept study to evaluate the anti-EBV activity of 4 grams of valomaciclovir (2 grams BID) for 21 days in subjects with infectious mononucleosis documented to be caused by primary EBV infection. Otherwise healthy subjects (≥15 years old) referred to us with a clinical diagnosis of primary infectious mononucleosis will be screened and those with laboratory-confirmed primary EBV infection will be enrolled.

DETAILED DESCRIPTION:
Subjects will be seen 2 times a week for 3 weeks and then weekly for 3 weeks. Clinical findings, clinical lab tests, EBV viral loads, and EBV antibody titers will be obtained at each clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 years or older
* Within 14 days of initial symptoms of present illness diagnosed by a health care provider as infectious mononucleosis and confirmed to be due to primary EBV by antibody profile. The criteria for antibody confirmation of primary EBV at the screening visit are: 1)Positive for anti-EBV VCA IgM antibody and negative for anti-EBV EBNA1 IgG antibody; 2)EBV antibody testing will be done in the Clinical Virology Research Laboratory using commercial ELISA kits (Diamedix Corporation, Miami, FL).
* Willingness to sign the Informed Consent Form (ICF)
* Willingness to contribute samples of blood and oral washings at regular intervals
* Males and females must use effective contraception during treatment and for at least 90 days following treatment
* Negative pregnancy test result at the Screening Visit for females of childbearing potential (including females who have had a bilateral tubal ligation). Female patients of childbearing potential must be willing to use an approved method of double-barrier contraception (hormonal plus barrier or barrier plus barrier, eg, diaphragm plus condom) from the time of first dose administration until 90 days after completion of dosing and male patients with female partners of childbearing potential must be willing to use a condom. Patients who are sterile or infertile (defined as those who are postmenopausal or have undergone a complete hysterectomy) are eligible.
* Estimated creatinine clearance (Cockcroft and Gault method) ≥ 60 ml/min
* Absolute neutrophil count ≥ 1000 cells/microliter
* Platelets ≥ 100,000/microliter
* Hemoglobin ≥ 9.5 g/dL

Exclusion Criteria:

* Previous history of infectious mononucleosis-like illness
* Immunosuppressed due to medical disease and/or immunosuppressive or immunomodulating medications (e.g., corticosteroids prior to enrollment, cytotoxic drugs, interferons)
* Another intercurrent viral infection (including HIV), based on history or referring physician medical evaluation
* More than 7 days elapsed since onset of illness (including screening time)
* The following concomitant medications are prohibited: probenecid, trimethoprim, myelosuppressive therapies, and medications known to be nephrotoxic
* Breast feeding during the study
* Corticosteroids are not permitted. If they are prescribed by the subject's primary physician for treatment of this acute disease after the subject has enrolled, the subject will be replaced.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry H Balfour, MD, Principal Investigator — Professor of Laboratory Medicine & Pathology, and Pediatrics
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Balfour HH Jr, Holman CJ, Hokanson KM, Lelonek MM, Giesbrecht JE, White DR, Schmeling DO, Webb CH, Cavert W, Wang DH, Brundage RC. A prospective clinical study of Epstein-Barr virus and host interactions during acute infectious mononucleosis. J Infect Dis. 2005 Nov 1;192(9):1505-12. doi: 10.1086/491740. Epub 2005 Sep 26. PMID 16206064
- [Background] Balfour HH Jr, Hokanson KM, Schacherer RM, Fietzer CM, Schmeling DO, Holman CJ, Vezina HE, Brundage RC. A virologic pilot study of valacyclovir in infectious mononucleosis. J Clin Virol. 2007 May;39(1):16-21. doi: 10.1016/j.jcv.2007.02.002. Epub 2007 Mar 21. PMID 17369082
- [Background] Rea TD, Russo JE, Katon W, Ashley RL, Buchwald DS. Prospective study of the natural history of infectious mononucleosis caused by Epstein-Barr virus. J Am Board Fam Pract. 2001 Jul-Aug;14(4):234-42. PMID 11458965
- [Background] Cameron B, Galbraith S, Zhang Y, Davenport T, Vollmer-Conna U, Wakefield D, Hickie I, Dunsmuir W, Whistler T, Vernon S, Reeves WC, Lloyd AR; Dubbo Infection Outcomes Study. Gene expression correlates of postinfective fatigue syndrome after infectious mononucleosis. J Infect Dis. 2007 Jul 1;196(1):56-66. doi: 10.1086/518614. Epub 2007 May 24. PMID 17538884
- [Background] Torre D, Tambini R. Acyclovir for treatment of infectious mononucleosis: a meta-analysis. Scand J Infect Dis. 1999;31(6):543-7. doi: 10.1080/00365549950164409. PMID 10680982
- [Background] Silins SL, Sherritt MA, Silleri JM, Cross SM, Elliott SL, Bharadwaj M, Le TT, Morrison LE, Khanna R, Moss DJ, Suhrbier A, Misko IS. Asymptomatic primary Epstein-Barr virus infection occurs in the absence of blood T-cell repertoire perturbations despite high levels of systemic viral load. Blood. 2001 Dec 15;98(13):3739-44. doi: 10.1182/blood.v98.13.3739. PMID 11739180
- [Background] Hislop AD, Taylor GS, Sauce D, Rickinson AB. Cellular responses to viral infection in humans: lessons from Epstein-Barr virus. Annu Rev Immunol. 2007;25:587-617. doi: 10.1146/annurev.immunol.25.022106.141553. PMID 17378764
- [Background] Hislop AD, Kuo M, Drake-Lee AB, Akbar AN, Bergler W, Hammerschmitt N, Khan N, Palendira U, Leese AM, Timms JM, Bell AI, Buckley CD, Rickinson AB. Tonsillar homing of Epstein-Barr virus-specific CD8+ T cells and the virus-host balance. J Clin Invest. 2005 Sep;115(9):2546-55. doi: 10.1172/JCI24810. Epub 2005 Aug 18. PMID 16110323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University of Minnesota students that contracted Mono and wsere seen at the student health center
Groups:
- Valomaciclovir: Valomaciclovir 2 grams orally twice daily for 21 days
  Valomaciclovir : 4 grams orally of valomaciclovir (2 grams BID) for 21 days.
- Placebo: placebo 2 tablets twice daily for 21 days
  placebo : Placebo tablets orally twice daily for 21 days.
Period: Overall Study
Arm/Group | Valomaciclovir | Placebo
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: College students infected with mono
Groups:
- Total: Total of all reporting groups
Arm/Group | Valomaciclovir | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Customized [Number; unit: particpants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Clinical Symptoms and Reductions in Viral Burden From Baseline
Description: All subjects had confirmed cases of EB and will be assessed for Improvement of clinical symptoms (ie: tiredness, nausea etc)and reduction in viral burden from baseline
Time Frame: 21 days
Measure: Number; unit: participants
Arm/Group | Valomaciclovir | Placebo
Number analyzed (Participants) | 12 | 11
participants | 12 | 11

2. Secondary Outcome: Number of Participants Who Experienced Adverse Events During the Study Safety and Tolerability
Description: Assessing adverse events in participants to see if this drug causes more or less side effects
Time Frame: 15 days
Measure: Number; unit: participants
Arm/Group | Valomaciclovir | Placebo
Number analyzed (Participants) | 12 | 11
participants | 12 | 11

ADVERSE EVENTS:
Arm/Group | Valomaciclovir | Placebo
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/11
Other Adverse Events (participants affected / at risk) | 7/12 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valomaciclovir (N=12) | Placebo (N=11)
Pancreatitis (Endocrine disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valomaciclovir (N=12) | Placebo (N=11)
Abdominal Pain (Gastrointestinal disorders) | 6 (6) | 5 (5)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Nausea (Gastrointestinal disorders) | 7 (7) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No